CLINICAL TRIAL: NCT03489980
Title: Influence of the Coloring of a Complex Form on Anxiety Associated With Care.
Acronym: COLORI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CHITS-06; 2017-A03537- 49 (Other: IdRCB)
Record Dates: First submitted 2018-03-20; First posted 2018-04-06 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Anxiety
Keywords: STAI Questionnaire; ECTM2-Qa
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ambulatory consultation waiting room: Patient from ambulatory consultation waiting room Group, coloring-type artistic task of a complex form before a medial consultation with hospital practitioner.
  Interventions: Other: coloring-type artistic task of a complex form
- Hemodialysis service: Patient from ambulatory consultation waiting room Group, coloring-type artistic task of a complex form during hemodialysis.
  Interventions: Other: coloring-type artistic task of a complex form
- Day hospitalization service : psychiatry: Patient from ambulatory consultation waiting room Group, coloring-type artistic task of a complex form during day hospitalization.
  Interventions: Other: coloring-type artistic task of a complex form

INTERVENTIONS:
Other: coloring-type artistic task of a complex form — coloring-type artistic task of a complex form

SUMMARY:
Evaluate the contribution of a coloring-type artistic task of a complex form in the reduction of anxiety related to care and pathology by a self-questionnaire "State-Trait anxiety inventory" and a self-questionnaire on the experience of the activity, in 3 different medical situations: in day hospitalization service in psychiatry, in hemodialysis service and in an ambulatory consultation waiting room.

DETAILED DESCRIPTION:
Evaluate the contribution of a coloring-type artistic task of a complex form in the reduction of anxiety related to care and pathology by a self-questionnaire "State-Trait anxiety inventory" and a self-questionnaire on the experience of the activity, in 3 different medical situations.

ELIGIBILITY:
Inclusion Criteria:

Psychiatric Day Hospital Group:

* Men or women over the age of 18 and under the age of 65.
* Admitted to psychiatric day hospital for at least 10 consecutive days of care.
* Person able to perform a coloring and answer a questionnaire, without severe deterioration of the general condition according to the assessment of the investigator.
* Patient with stabilized schizophrenia (F20.0).

Hemodialysis Service Group:

* Men or women over the age of 18 and under the age of 65.
* Person able to perform a coloring and answer a questionnaire, without severe deterioration of the general condition according to the assessment of the investigator.
* Person having had at least 6 hemodialysis sessions.
* Valid dominant arm (allowing coloring - no fistula).
* Person currently on dialysis treatment.

Group Ambulatory consultation waiting room:

* Men or women over the age of 18 and under the age of 65.
* Person able to perform a coloring and answer a questionnaire, without severe deterioration of the general condition according to the assessment of the investigator.
* Consultant a practitioner at the hospital.

Exclusion Criteria:

* Person with advanced cognitive impairment that alters the questionnaire response or coloring as assessed by the investigator.
* Opposition of the volunteer.
* No affiliation to a social security scheme (beneficiary or beneficiary).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient from Sainte-Musse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Change in anxiety state | 20 minutes
  Self questionnaire STAI-YA before and after coloring

SECONDARY OUTCOMES:
Anxiety trait | 0 minutes
  Self questionnaire STAI-YB
Experience of activity | 10 minutes
  Self questionnaire ECTM-Q2a after coloring

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Knefati, MD, Study Director — Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer
Locations (1):
- Centre hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dias Alves M, Olmi E, Durand JY, Mitri F, Knefati Y, Vion-Dury J. Coloring complex shapes decreases patient anxiety in three care environments: a pilot study with color analysis. Front Psychol. 2024 Feb 21;15:1336202. doi: 10.3389/fpsyg.2024.1336202. eCollection 2024. PMID 38449752